CLINICAL TRIAL: NCT04616118
Title: Comparing Modes of Telehealth Delivery:Phone vs. Video Visits
Brief Title: Comparing Modes of Telehealth Delivery: Phone vs. Video Visits (ASSIST)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Maria Danila, MD, MSc, MSPH, Associate Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB-300005184
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Rheumatic Disease; Cardiac Disease; Primary Care; Infectious Disease
MeSH Terms: conditions — Rheumatic Diseases; Heart Diseases; Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phone (Experimental): Participants randomized to this arm will receive usual care via telephone only
  Interventions: Other: Phone Visit
- Video (Experimental): Participants randomized to this arm will receive usual care via video call
  Interventions: Other: Video Visit

INTERVENTIONS:
Other: Phone Visit — Participants randomized to this arm will receive usual care via telephone only
  Arms: Phone
Other: Video Visit — Participants randomized to this arm will receive usual care via video call
  Arms: Video

SUMMARY:
Given the current public health crisis the use of telehealth consultation visits including phone-only and video visits has exponentially increased. This study will investigate if the conduct of telehealth phone only visits is non-inferior in terms of patient satisfaction/experience, adherence to post-visit recommendations such as medications, blood work and other medical testing, follow up care, when compared to the conduct of video delivered telehealth visits. Patients will be randomized to receive a routine care visit via phone only vs. video.

DETAILED DESCRIPTION:
Telemedicine and an emerging field of novel care delivery modalities, which encompasses all forms of remote-based care. These include asynchronous (store-and-forward) and consultative care by specialists, mobile-device based care, and real-time video chat, and synchronous telemedicine. Health care services delivered remotely through telecommunications and video technology is steadily increasing as technology evolves and access becomes more widely available. The increasing availability of personal technology - 89% Americans have internet access, 77% are online daily - offers patients and clinicians the opportunity to utilize real-time virtual communication to enhance access for patients when transportation challenges, schedules, or physical disability make office visits difficult in any geography. With the increased use of technology in healthcare, much emphasis has been placed on telemedicine as it can extend the services of providers to remote locations and overcome the barrier of proximity. This expands access to care and has the potential of making healthcare services more convenient for many patients who otherwise might suffer access barriers.

It is increasingly evident that telehealth can improve access to healthcare services and specialists; prevent unnecessary delays in receiving care, and facilitate coordinated care and interprofessional collaboration. The World Health Organization affirms the efficacy of telehealth as an effective service delivery model for professionals.

Telemedicine has been shown to improve health outcomes, increase communication with providers, increase access to high-quality service, decrease travel time, decrease missed appointments, decrease wait time, decrease repeat admissions, increase self-awareness, increase medication adherence, and increase self-monitoring of chronic conditions. The technical quality of telehealth consultation (e.g. audio and visual quality of a videoconference) has been shown to influence clinicians' willingness to practice in this manner and the satisfaction of users. A recent systematic review on patient satisfaction with telemedicine found that patient satisfaction can be associated with the modality of telehealth, but factors of effectiveness and efficiency are mixed. Telehealth is a feasible option to expand practices to remote areas without having to relocate or expand. Understanding the perceived relative value of different modes of healthcare services may help to shape the use of virtual or remote healthcare technologies. System learning that demonstrates the value of different types of "visits" for the system and the patient is essential.

ELIGIBILITY:
Inclusion Criteria:

* Access to a phone and video call capacity
* A minimum of 1 visits in the last year with their provider
* Medicare/Medicaid eligible

Exclusion Criteria:

•Individuals not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | 36 hours post visit
  Patient satisfaction with type of visit. Satisfaction will be measured using the 11-point ARHQ-CAHPS patient satisfaction instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Danila, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donelan K, Barreto EA, Sossong S, Michael C, Estrada JJ, Cohen AB, Wozniak J, Schwamm LH. Patient and clinician experiences with telehealth for patient follow-up care. Am J Manag Care. 2019 Jan;25(1):40-44. PMID 30667610
- [Background] Wade V, Smith AC. Research methods and methodology in telemedicine. J Telemed Telecare. 2017 Oct;23(9):757-758. doi: 10.1177/1357633X17733088. No abstract available. PMID 29070002
- [Background] Batsis JA, Pletcher SN, Stahl JE. Telemedicine and primary care obesity management in rural areas - innovative approach for older adults? BMC Geriatr. 2017 Jan 5;17(1):6. doi: 10.1186/s12877-016-0396-x. PMID 28056832
- [Background] Wade VA, Eliott JA, Hiller JE. Clinician acceptance is the key factor for sustainable telehealth services. Qual Health Res. 2014 May;24(5):682-94. doi: 10.1177/1049732314528809. Epub 2014 Mar 31. PMID 24685708
- [Background] Kruse CS, Soma M, Pulluri D, Nemali NT, Brooks M. The effectiveness of telemedicine in the management of chronic heart disease - a systematic review. JRSM Open. 2017 Feb 1;8(3):2054270416681747. doi: 10.1177/2054270416681747. eCollection 2017 Mar. PMID 28321319